CLINICAL TRIAL: NCT01837745
Title: Differentiated Thyroid Cancer: is There a Need for Radioiodine Ablation in Low Risk Patients?
Acronym: ESTIMABL2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-A01569-34; 2012/1913 (Other: CSET number)
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Low Risk Differentiated Thyroid Cancer
MeSH Terms: interventions — Thyrotropin Alfa; Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation group (Active Comparator): * Administration of 1.1 GBq of I131 is given after the second intramuscular injections of rhTSH (0.9 mg). A whole body scan (WBS) is performed 2 to 5 days after the administration or I131 with determination of the neck uptake.
  * Follow-up consists in:
    * 10 (+/- 2 months) after randomization: neck ultrasound + a serum Tg measurement after rhTSH stimulation
    * 2 years (+/- 2 months) after randomization: serum Tg measurement under LT4 treatment (Tg/LT4)
    * 3 years (+/- 2 months) after randomization: neck ultrasound and a serum Tg/LT4
    * 4 years (+/- 2 months) after randomization: a serum Tg/LT4
    * 5 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
    * 8 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
    * 10 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
    * 12 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
  Interventions: Drug: rhTSH stimulation; Drug: I131; Other: Follow up
- Follow up group (Experimental): Patients randomized in the follow up group neither received 131I nor rhTSH. Patients will undergo the same followup procedures as patients randomized to the ablation group, except that at 10 months after randomization, Tg will be measured under LT4 treatment and not after rhTSH stimulation.
  Interventions: Other: Follow up

INTERVENTIONS:
Drug: rhTSH stimulation — Intramuscular injections of rhTSH (0.9 mg) on two consecutive days on LT4 treatment
  Other Names: Thyrogen
  Arms: Ablation group
Drug: I131 — An activity of 1.1 GBq of I131 is given orally 24 hours after the second injection of rhTSH.
  Arms: Ablation group
Other: Follow up — * 10 (+/- 2 months) after randomization: a neck ultrasound and a serum Tg measurement after rhTSH or LT4 stimulation
  * 2 years (+/- 2 months) after randomization: a serum Tg measurement under LT4 treatment (Tg/LT4)
  * 3 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
  * 4 years (+/- 2 months) after randomization: a serum Tg/LT4
  * 5 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
  * 8 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
  * 10 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4
  * 12 years (+/- 2 months) after randomization: a neck ultrasound and a serum Tg/LT4

SUMMARY:
Open-label randomized phase III trial, using a non-inferiority comparison design. After randomization,patients will receive either post-operative radioiodine ablation with an activity of 1.1 GBq (30 mCi) after stimulation by rhTSH, and then be followed-up (ablation group) or be followed-up (without postoperative radioiodine ablation) (follow-up group).

The objective is to assess the non-inferiority of the proportion of patients without tumor-related event evaluated at three years after randomisation in the absence of radioiodine ablation (follow-up group) compared to the ablation group, in patients with low-risk differentiated thyroid cancer treated with total thyroidectomy with or without lymph node dissection (pT1am N0 or Nx, pT1b N0 or Nx)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with differentiated thyroid cancer (papillary, follicular or with Hurthle cells) in the absence of aggressive histological subtypes (poorly differentiated, tall-clear-cylindric cell, diffuse sclerosing or with an anaplastic component)
2. Patients having undergone a total thyroidectomy with complete (R0) tumor resection, with or without lymph node neck dissection
3. Total thyroidectomy performed 2 to 5 months before inclusion
4. Patients with low risk of recurrence: pT1amN0 or pT1amNx with a sum of the size of the lesions above 1 cm and equal to or less than 2 cm, or pT1bN0 or pT1bNx (TNM 2010 classification).
5. Post-operative neck ultrasound (performed 2 to 5 months after surgery) showing the absence of abnormalities in the lateral lymph node compartments, or if abnormalities, no lymph nodes with abnormal cytology and/or thyroglobulin concentration in the aspirate fluid > 10 ng/mL
6. Age >=18 years
7. Performance status of 0 or 1
8. Patients who signed the informed consent
9. Patients who can be followed-up annually during 5 years in order to assess the objectives of the study
10. Women of childbearing age should have a negative pregnancy test before any radioiodine administration
11. Both patients with or without thyroglobulin antibodies are eligible

Exclusion Criteria:

1. Patients having undergone less than a total thyroidectomy
2. Patients with aggressive histotype (poorly differentiated, tall-clear-cylindric cell, diffuse sclerosing, or with an anaplastic component)
3. Patients having undergone total thyroidectomy less than 2 months or more than 5 months before inclusion
4. Patients with cancer classified as pT1a unifocal (in which ablation is not necessary), or pT1N1, pT2, pT3, pT4 or N1 (who have a higher risk of recurrence) (classification TNM 2010)
5. Patient with known distant metastasis
6. Abnormal post-operative neck ultrasound of the lateral lymph node compartments
7. Patients with another malignancy not in remission for at least 2 years (except for in situ cervix uterine cancer, basocellular skin cancer)
8. Patients with a recent history of drugs affecting thyroid function, including injection of radiocontrast agents during the last 8 weeks.
9. Patients previously treated with radioactive iodine or who previously underwent a whole body scan with radioactive iodine
10. Pregnant or breast feeding women
11. Subject with any kind of disorder that may compromise his/her ability to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patient without event at 3 years following randomization | assessed up to 3 years

SECONDARY OUTCOMES:
Lachrymal and Salivary Glands Toxicities | Assessed up at baseline, 2 months, 10 months and 3 years after randomization
Patient's quality of life, anxiety and fear of recurrence | at inclusion, 2 months after inclusion, 10 months and 3 years after randomization
Rate of patients without event | at 5 years following randomization
Rate of events adjusted on the initial lymph node status | at 3 and 5 years following randomization
Recurrence rate (histologically proven) | at 3 years following randomization and then at 5 years
Rate of cure after an event | at 5 years after randomization
Cost of treatment and follow-up | at 3 years after randomization
Rate of events adjusted on tumoral molecular characterization | 3 and 5 years after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Leboulleux S, Bournaud C, Chougnet CN, Lamartina L, Zerdoud S, Do Cao C, Catargi B, Dygai I, Kelly A, Barge ML, Vera P, Rusu D, Schneegans O, Roux J, Raymond P, Benisvy D, Eberle MC, Bidault S, Nascimento C, Bastie D, Giraudet AL, Bardet S, Le Moullec N, Roudaut N, Drui D, Godbert Y, Zalzali M, Drutel A, Morel O, Velayoudom FL, Al Ghuzlan A, Schlumberger M, Buffet C, Borget I. Thyroidectomy without radioiodine in patients with low-risk thyroid cancer: 5 years of follow-up of the prospective randomised ESTIMABL2 trial. Lancet Diabetes Endocrinol. 2025 Jan;13(1):38-46. doi: 10.1016/S2213-8587(24)00276-6. Epub 2024 Nov 22. PMID 39586309
- [Derived] Leboulleux S, Bournaud C, Chougnet CN, Zerdoud S, Al Ghuzlan A, Catargi B, Do Cao C, Kelly A, Barge ML, Lacroix L, Dygai I, Vera P, Rusu D, Schneegans O, Benisvy D, Klein M, Roux J, Eberle MC, Bastie D, Nascimento C, Giraudet AL, Le Moullec N, Bardet S, Drui D, Roudaut N, Godbert Y, Morel O, Drutel A, Lamartina L, Schvartz C, Velayoudom FL, Schlumberger MJ, Leenhardt L, Borget I. Thyroidectomy without Radioiodine in Patients with Low-Risk Thyroid Cancer. N Engl J Med. 2022 Mar 10;386(10):923-932. doi: 10.1056/NEJMoa2111953. PMID 35263518